CLINICAL TRIAL: NCT04818541
Title: Early Feasibility Study of the Vivasure PerQseal® Closure Device System After Use of the Impella Device for Cardiogenic Shock or Protected Percutaneous Coronary Intervention
Brief Title: PerQseal® Impella Early Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivasure Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P849-00
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Percutaneous Large Hole Vascular Closure
Keywords: vascular closure; arterial closure; vascular closure device; large hole percutaneous closure; large bore percutaneous closure

STUDY DESIGN:
Intervention Model Description: Early Feasibility Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Protected Percutaneous Coronary Intervention (Experimental): Subjects with a femoral arteriotomy created with 13 to 14 F sheaths (arteriotomy up to approximately 18 F) and in whom an Impella device was used for PPCI. Duration of Impella use ≤ 6 hours if used for PPCI.
  Interventions: Device: PPCI
- Cardiogenic shock (Experimental): Subjects with a femoral arteriotomy created with 13 to 14 F sheaths (arteriotomy up to approximately 18 F) and in whom an Impella device was used for cardiogenic shock. Duration of Impella use > 8 hours and ≤ 4 days.
  Interventions: Device: Cardiogenic shock

INTERVENTIONS:
Device: PPCI — Closure of the femoral access site with PerQseal device at the end of the PPCI index procedure and removal of the Impella pump.
  Other Names: Percutaneous PerQseal device closure
  Arms: Protected Percutaneous Coronary Intervention
Device: Cardiogenic shock — Closure of the femoral access site with PerQseal device after removal of the Impella pump.
  Other Names: Percutaneous PerQseal device closure
  Arms: Cardiogenic shock

SUMMARY:
The purpose of this Clinical Investigation Plan is to assess the initial feasibility results of the PerQseal® device, when used on this very specific Impella population. Safety and effectiveness will be assessed in patients where an Impella device was used for either cardiogenic shock or PPCI. Closure of femoral arterial access sites created with 13 to 14 F sheaths will be studied, assessing the need for alternative therapy other than manual compression or adjunctive endovascular ballooning.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, single arm EFS. Patients undergoing use of an Impella device for cardiogenic shock or PPCI, requiring an arteriotomy created by 13 to 14 F sheaths (arteriotomies up to approx. 18 F), via the common femoral artery will be screened against the study inclusion/exclusion criteria. If the patient meets study eligibility requirements, they shall be invited to participate, provide informed consent, and shall subsequently be assigned a study ID number. Enrollment will occur at the point where the PerQseal study device first enters the patient's body.

The planned enrollment is a minimum of 20 treated patients at a maximum of 5 study sites located in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years,
2. Use of an Impella CP or 2.5 Impella device via the common femoral artery for protected percutaneous coronary intervention (PPCI) or cardiogenic shock,
3. Duration of Impella use > 8 hours and ≤ 4 days if used for cardiogenic shock
4. Duration of Impella use ≤ 6 hours if used for PPCI.
5. Impella access sheath between 13 and 14 F,
6. Potential subject or authorized representative willing and able to provide appropriate study-specific informed consent,
7. Females who are not pregnant or lactating and not planning to become pregnant for the duration of the study.

Baseline Exclusion Criteria:

1. Evidence of systemic bacterial or cutaneous infection, including groin infection,
2. Known bleeding diathesis, definite or potential coagulopathy, platelet count < 100,000/µl or subjects on long term anticoagulants with an INR > 2 within 12 hours prior to index procedure,
3. Significant anemia (hemoglobin <9 g/dL or hematocrit < 27%), within 24 hours prior to index procedure,
4. Known type II heparin-induced thrombocytopenia,
5. Unilateral or bilateral lower extremity amputation.
6. Rest pain (e.g., Rutherford category 4 or greater), documented untreated iliac or common femoral artery diameter stenosis > 50% or previous bypass surgery/stent placement in the common femoral artery of target leg,
7. Known existing nerve damage in the target leg,
8. Known allergy to any of the materials used in the PerQseal® device (refer to Instructions for Use),
9. Subject unsuitable for surgical repair of the target leg access site,
10. Subject has undergone a percutaneous procedure greater than 8 F sheath in the target leg, within the 90 days prior to index procedure,
11. Subject has undergone a percutaneous procedure of 8 F sheath or less using an absorbable or suture mediated closure device for hemostasis, in the target vessel, within the 90 days prior to index procedure,
12. Prior evidence of anterior calcification within 10 mm proximal or distal to arteriotomy site,
13. Target femoral artery diameter is less than 6 mm in diameter,
14. Subject is enrolled in another investigational medical device or drug study which has not completed the required primary endpoint follow-up,
15. Subject has been previously enrolled in this clinical study.
16. Current COVID-19 infection (with or without symptoms), recent positive test for COVID-19, or recent exposure to a person with COVID-19 infection.

Procedural Exclusion Criteria:

1. Initial common femoral arterial access achieved with manual palpation or blind arterial stick access, without use of an image guided approach (ultrasound or angiography).
2. Difficult dilation during initial target femoral artery access (e.g., that damages or kinks sheath dilators) while step-dilating up to the large-bore device,
3. During arterial puncture, the target femoral artery suspected to have experienced a back arterial wall needle puncture or underwent > one needle puncture during the primary procedure,with a needle larger than a Micropuncture needle (18 gauge)
4. Subject has a tissue tract (i.e., estimated distance from skin entry point to arterial anterior surface at arteriotomy) expected to be greater than 8 cm,
5. Significant blood loss/transfusion (defined as requiring transfusion of 4 or more units of blood products) during primary procedure or within 30 days prior to index procedure,
6. Activated clotting time (ACT) > 300 seconds immediately prior to sheath removal or if ACT measurements are expected to be > 300 seconds for more than 24 hours after index procedure,
7. Target puncture site is in a vascular graft,
8. Target arteriotomy in the profunda femoris or superficial femoral artery or is in common femoral artery, but within 10 mm proximal of the bifurcation of the superficial femoral/ profunda femoris artery,
9. Target arteriotomy located above the inferior epigastric artery and/or above the inguinal ligament based on bony landmarks,
10. Subjects with an acute hematoma > 4 cm diameter, arteriovenous fistula, pseudoaneurysm, or intraluminal thrombosis at the target access site,
11. Evidence of bleeding around the Impella sheath (BARC type 2 or higher),
12. Angiographic evidence of arterial laceration, dissection or stenosis within the femoral artery that would preclude use of the PerQseal® device,
13. Uncontrolled hypertension (systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg) just prior to planned vascular closure.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Safety: Major Access Site Complications | through 30 days
  The primary safety endpoint is the rate of major access site complications attributable to the PerQseal® device. As per FDA definitions for Major access site complications.
Efficacy: Time to Hemostasis | 20 minutes
  Elapsed time in minutes from PerQseal® Introducer sheath removal to first observed cessation of common femoral artery (CFA) bleeding (excluding cutaneous or subcutaneous oozing, and in the absence of a developing hematoma).

SECONDARY OUTCOMES:
Safety: Incidence of Minor Access Site Complications | through 30 days
  Incidence and severity of minor access site complications attributable to the PerQseal® device, adapted from FDA-provided definitions.
Efficacy: PerQseal® Device Technical Success Rate | 10 minutes
  PerQseal® Device Technical Success Rate, defined as the number of PerQseal® devices that are deployed and achieve hemostasis (i.e., cessation of bleeding (excluding cutaneous or subcutaneous oozing)) without need for firm, adjunctive manual compression for greater than 10 minutes or alternative treatment (other than adjunctive endovascular ballooning) at target access site, divided by the total number of PerQseal® devices where deployment was attempted.
Efficacy: PerQseal® Treatment Success Rate | through 30 days
  PerQseal® Treatment Success Rate, defined as the number of subjects who meet PerQseal® Device Technical Success without experiencing a Major Access Site Complication, divided by the total number of subjects where PerQseal® device deployment was attempted.
Efficacy: Time to Device Deployment | 20 minutes
  Time to Device Deployment, defined as the time from insertion of the PerQseal® device into the PerQseal Introducer sheath to complete removal of the PerQseal® device delivery system and PerQseal® Introducer sheath from the subject following PerQseal® deployment.
Efficacy: Overall Procedural Time | 4 days
  Overall Procedural Time, defined as the time from first invasive contact with the subject's groin to completion of all aseptic procedures related to the groin and index procedure.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - The Valley Hospital, Ridgewood, New Jersey
  - University of Buffalo, Buffalo, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No